CLINICAL TRIAL: NCT06847152
Title: Spatial Memory and Temporal Lobe Epilepsy
Acronym: EPINAVIG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHMS24007
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy Lobe Temporal; Healthy; Epilepsy
Keywords: epilespsy; lobe temporal; spatial memory; navigation task; accelerated forgetting
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy participant (Experimental): spatial memory test to healthy participant
  Interventions: Diagnostic Test: spatial memory test
- Epileptic patient (Experimental): spatial memory test to epileptic patient
  Interventions: Diagnostic Test: spatial memory test

INTERVENTIONS:
Diagnostic Test: spatial memory test — The assessment of spatial memory corresponds in our study to a navigation task, i.e. learning a route through the hospital. The route encoding phase is first carried out. The participant follows the experimenter, with the instruction to pay close attention to the route in order to be able to do it again alone. For directions, it is said "this way" or "that way" and not "left" or "right". The route includes 18 intersections.
  The participant immediately does the route again alone. The number of correct answers (BR), i.e. correct directions taken at each intersection, is counted as well as the time to complete the route (TR). Direction errors are corrected. This is recall 1.
  The participant is then asked to do the route a second time. The correct answers and the times to complete the route are recorded. Errors are corrected (feedback). This is recall 2.
  If the participant makes a mistake on recall 1 or 2, a third attempt is made. This is recall 3.
  After an interval of 1 hour, the partic

SUMMARY:
Temporal lobe epilepsy (TLE) can cause memory disorders, including long-term forgetfulness due to a failure to consolidate verbal but also spatial information. The forgetting phenomenon presented by these epileptic patients is called accelerated forgetting in the literature and remains difficult to objectify during cognitive assessments. It is indeed particularly complicated to evaluate long-term spatial memory and to account for the topographical complaint, although recurrent, of patients with this TLE.

A navigation task being proposed as part of the neuropsychological assessment of patients with a spatial memory complaint, it is interesting to study the performance pattern of patients with TLE by comparing them to a group of control subjects matched in age and gender in order to verify whether there is significant long-term forgetting and whether there is a significant difference between Right TLE and Left TLE. Indeed, several studies have demonstrated this accelerated long-term forgetting in epileptic patients (Cassel et al., 2016; Lemesle et al., 2017; Landry et al., 2022; Blake et al., 2020) but few with a retention delay of several weeks (Tramoni et al., 2009). This study allows us to statistically analyze the effects of these two groups: epileptic patients and healthy volunteers, but also to combine the effect of the laterality of epilepsy specifically on spatial memory performance.

DETAILED DESCRIPTION:
In order to assess the long-term spatial memory capacities of epileptic patients with memory complaints, a navigation task was proposed as part of the neuropsychological assessment. This task corresponds to learning a route within the hospital. It is composed of a learning phase and then the patient is asked to repeat the route one hour later and then six weeks later, in order to check for the presence or absence of long-term forgetting. We wanted to study the results of patients with temporal lobe epilepsy (TLE) by comparing them to a group of healthy volunteers matched in age and gender in order to check whether there is significant long-term forgetting and whether there is a significant difference between Right TLE and Left TLE. This study therefore aims to statistically analyze the effects of these two groups: epileptic patients and healthy volunteers, but also to combine the effect of the laterality of epilepsy specifically on spatial memory performance. It will also be interesting to observe whether there is a difference between men and women in the healthy volunteer group for spatial memory learning.

ELIGIBILITY:
Inclusion Criteria:

- healthy volunteers meeting each of the following criteria:

* Aged over 18 years
* Right-handed*
* Free of known neurological pathology
* Signed consent
* Matched in age (+ or - 5 years) and gender with epileptic patients presenting the characteristics below:

  * Right-handed*
  * adult
  * presenting temporal lobe epilepsy, whose lateralization of the epileptogenic focus (right or left) has been objectified by an examination (EEG and/or MRI),
  * having carried out a neuropsychological assessment including the navigation task,
  * having been informed of the study, and consenting to the processing of their data

Exclusion Criteria:

* Person referred to in Article L1121-5 of the Public Health Code: Pregnant, parturient, or breastfeeding women
* Person referred to in Article L1121-6 of the Public Health Code: persons deprived of their judicial or administrative freedom
* Person referred to in Article L1121-8 of the Public Health Code: persons subject to a legal protection measure or unable to express their consent
* Person referred to in Article L1121-8-1 of the Public Health Code: persons not affiliated to a social security scheme
* Left-handed participants
* Participants familiar with the premises of the Centre Hospitalier Métropole Savoie
* Not speaking French

Exclusion criteria

Patients who have undergone epilepsy neurosurgery between the initial visit and the secondary visit of the neuropsychological assessment will not be paired with a healthy volunteer. Their data will not be studied.

Volunteers whose pretest scores reveal a cognitive disorder (pathological threshold > 1.65) will not perform the navigation task. They will then be referred to a neurologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
Changes of the number of correct responses from 1h to 6 weeks, compared between healthy volunteers and epileptic patients | 1 hour and 6 weeks
  The number of correct responses is defined as the number of intersections correctly crossed.

SECONDARY OUTCOMES:
Changes in test performance from 1h to 6 weeks, compared according to epileptogenic focus (right or left) lateralization. | at 1 hour and 6 weeks.
  Test performance is evaluated by completion time (TR) and number of correct responses (BR).
Changes in test performance from 1h to 6 weeks, compared between male and female in the healthy volunteers group | at 1 hour and 6 weeks.
  Test performance is evaluated by completion time (TR) and number of correct responses (BR).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Métropole Savoie, Chambéry, Savoie, France

IPD SHARING:
Plan to Share IPD: No